CLINICAL TRIAL: NCT07003230
Title: Effect of Vegan Diet on Microbiome and Metabolism
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Liu Zhanguo, Professor, Zhujiang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 32271230
Record Dates: First submitted 2025-05-08; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Vegan Diet
MeSH Terms: interventions — Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effect of vegan diet on microbiome and metabolism (Experimental)
  Interventions: Dietary Supplement: vegan and omnivorous diet

INTERVENTIONS:
Dietary Supplement: vegan and omnivorous diet — Participants underwent a 2-week omnivorous diet intervention, followed by a 2-week vegan diet intervention

SUMMARY:
The goal of this interventional study is to investigate how vegan diet affects health in healthy volunteers, Men and women ages 20 - 30 years old. The main questions it aims to answer are:

Change in Microbial community composition and metabolic alterations Changes in plasma metabolic profile. Researchers will compare changes in microbiota and plasma metabolites profile to see the influence of vegan diet in health. In the dietary trial, participants were first assigned to a 2-week omnivorous diet phase, then switched to a 2-week vegetarian diet phase

ELIGIBILITY:
Inclusion Criteria: healthe Participants, ages 20-30 years old

Exclusion Criteria:

1. Oral antibiotic use or acute/chronic inflammation within the past 3 months;
2. Hormone intake within the past 3 months;
3. Use of any known interfering medications (e.g., insulin, glibenclamide, indomethacin, phentolamine, furosemide, phenytoin sodium, cortisone, etc.) or probiotics within the past month that may affect glucose or lipid metabolism;
4. Smoking or alcohol consumption;
5. Uncontrolled mental disorders (including a history of psychiatric hospitalization);
6. Currently participating in a weight loss or weight management program;
7. Following a special or medically prescribed diet (e.g., for celiac disease);
8. Comorbid cardiac or renal insufficiency;
9. Chronic constipation;
10. Hypertension;
11. Diabetes mellitus.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota composition in twenty participants | 14days，28days
  16S rDNA sequencing technology was used to identify the structural and functional changes of intestinal microbiota before and after vegan diet.

SECONDARY OUTCOMES:
Metabolomic profile of twenty participants in serum and feces | 14days, 28days
  To determine changes of the metabolomic profile in feces and serum after vegan diet

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Link VM, Subramanian P, Cheung F, Han KL, Stacy A, Chi L, Sellers BA, Koroleva G, Courville AB, Mistry S, Burns A, Apps R, Hall KD, Belkaid Y. Differential peripheral immune signatures elicited by vegan versus ketogenic diets in humans. Nat Med. 2024 Feb;30(2):560-572. doi: 10.1038/s41591-023-02761-2. Epub 2024 Jan 30. Erratum In: Nat Med. 2024 Jun;30(6):1785. doi: 10.1038/s41591-024-02884-0. PMID 38291301